CLINICAL TRIAL: NCT00137436
Title: A Phase 1/2 Safety And Pharmacokinetic Study Of SU011248 In Combination With Docetaxel (Taxotere) And Prednisone In Patients With Metastatic Hormone Refractory Prostate Cancer (HRPC)
Brief Title: Study Of SU011248 In Combination With Docetaxel (Taxotere) And Prednisone In Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181043
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Prostatic Neoplasms
Keywords: First-line treatment of metastatic hormone-refractory prostate cancer SUTENT in combination with docetaxel and prednisone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Sunitinib; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): SU011248 in combination with docetaxel and prednisone
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: SU011248

INTERVENTIONS:
Drug: Docetaxel — Docetaxel Phase 1 - escalating doses (60 and 75 mg/m2), intravenous therapy (IV), administered every 3 weeks. Phase 2 - Phase 1 optimal combination dose (75 mg/m2, IV, every 3 weeks).
  Other Names: Taxotere; Sunitinib malate; SUTENT
Drug: Prednisone — Prednisone Phase1/2 - 5 mg twice a day (BID), oral.
Drug: SU011248 — SU011248 Phase 1 - escalating doses (12.5, 37.5, and 50 mg), oral, administered on a 2-weeks on, 1-week off daily regimen (Schedule 2/1). Phase 2 - Phase 1 optimal combination dose (37.5 mg/day, oral, Schedule 2/1).

SUMMARY:
This is a multi-center, open-label, Phase 1/2 study of SU011248 (sunitinib malate, SUTENT) in combination with docetaxel and prednisone for the first-line treatment of metastatic hormone-refractory prostate cancer (mHRPC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Patients must have progressive hormone-refractory prostate cancer (HRPC): patients must have undergone primary hormone treatment (e.g. orchiectomy or gonadotropin releasing hormone analog with or without antiandrogens). For patients who received antiandrogen therapy, disease progression must have been determined after antiandrogen discontinuation
* Progressive disease based on either non-measurable disease and an elevated PSA OR measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Prior thalidomide, anti-vascular endothelial growth factor (VEGF) therapy, VEGF receptor inhibitor, platelet-derived growth factor (PDGF) receptor inhibitor or anti-angiogenic treatment of any kind including investigational therapy
* Prior chemotherapy
* Uncontrolled pain at baseline, impending complication from bone metastasis (fracture and/or compression) and/or presence of urinary obstruction (urinary retention, hydronephrosis)
* History of cardiac dysfunction, QT interval corrected for heart rate (QTc) >450 msec
* Central Nervous System (CNS) involvement

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2005-10; Primary Completion 2008-05 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (20):
  - Pfizer Investigational Site, Harvey, Illinois
  - Pfizer Investigational Site, Tinley Park, Illinois
  - Pfizer Investigational Site, Hobart, Indiana
  - Pfizer Investigational Site, Munster, Indiana
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Myrtle Beach, South Carolina
  - Pfizer Investigational Site, Clarksville, Tennessee
  - Pfizer Investigational Site, Franklin, Tennessee
  - Pfizer Investigational Site, Gallarin, Tennessee
  - Pfizer Investigational Site, Hermitage, Tennessee
  - Pfizer Investigational Site, Lebanon, Tennessee
  - Pfizer Investigational Site, Murfreesboro, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Smithville, Tennessee
  - Pfizer Investigational Site, Smyrna, Tennessee
  - Pfizer Investigational Site, Tullahoma, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Madison, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181043&StudyName=Study%20Of%20SU011248%20In%20Combination%20With%20Docetaxel%20%28Taxotere%29%20And%20Prednisone%20In%20Patients%20With%20Prostate%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Once the Optimal Combination Dose of SU011248, Docetaxel, and prednisone was determined in Phase 1, the study proceeded to Phase 2. There were 38 participants in Phase 1; those participants did not continue into Phase 2. Per FDAAA, only Phase 2 data are posted; timeframes are relative to Phase 2.
Groups:
- SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg: Sunitinib 37.5 milligrams (mg) plus (+) Docetaxel 75 mg per meters squared (mg/m^2) + Prednisone 5 mg given twice daily
Period: Overall Study
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Started | 55 (Phase 2 did not include 38 participants from Phase 1.)
Completed | 12
Not Completed | 43
Not completed — Adverse Event | 13
Not completed — Death | 2
Not completed — Lack of Efficacy | 17
Not completed — Withdrawal by Subject | 6
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Groups:
- SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg: SU011248 (Sunitinib Malate) 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg given twice daily
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 65.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Prostate Specific Antigen (PSA) Response
Description: PSA response rate, which is defined as a greater than or equal to a 50% decrease in PSA from baseline, that is subsequently confirmed.
Time Frame: Baseline, Day 1 of each 21-day cycle
Population: The intent-to-treat (ITT) population was defined as all patients enrolled in the study that receive at least 1 dose of study medication (SU011248 or docetaxel)
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 55
percentage of participants | 56.4 [42.3 to 69.7]

2. Secondary Outcome: Time to PSA Progression
Description: Defined as the time from start of study treatment to first documentation of PSA progression using the PSA Working Group criteria calculated as (first event date - first dose date + 1)/7. PSA progression is defined for patients with a PSA response, as a 50% increase over nadir (lowest) and increase in absolute-value PSA level by at least 5 nanograms per milliliter (ng/mL) [or back to baseline] and for patients without a PSA response as a 25% increase over baseline [or nadir (lowest)] and increase in absolute-value PSA level by at least 5 ng/mL, both confirmed by a second value.
Time Frame: Baseline to first documentation of PSA progression up to 28 days after date of last dose
Population: ITT
Measure: Median (Full Range); unit: weeks
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 55
weeks | 42.1 [33.1 to NA] — upper range not reached; the data was not mature.

3. Secondary Outcome: Duration of PSA Response (DPR)
Description: Defined as time from first documentation of PSA response (≥50% decrease in PSA from baseline that is subsequently confirmed) to first documentation of PSA progression (defined for patients with a PSA response as a 50% increase over nadir [lowest] and increase in absolute-value PSA level by at least 5 ng/mL [or back to baseline] and for patients without a PSA response as a 25% increase over baseline [or nadir / lowest] and increase in absolute-value PSA level by at least 5 ng/mL, both confirmed by a second value). Calculated as (end date for DPR - first PSA response + 1)/7.
Time Frame: Baseline to first documentation of PSA progression up to 28 days after date of last dose
Population: ITT; DPR only calculated for the subgroup of patients with PSA response rate.
Measure: Median (Full Range); unit: weeks
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 31
weeks | 39.1 [36.0 to NA] — upper range not reached; the data was not mature.

4. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR)
Description: Defined as confirmed complete response (CR: disappearance of all target lesions) or confirmed partial response (PR: ≥30% decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD) according to response evaluation criteria in solid tumors (RECIST). Confirmed responses are those that persist on repeat imaging study ≥4 weeks after initial documentation of response.
Time Frame: Baseline to first documentation of PSA progression up to 28 days after date of last dose
Population: ITT; N=participants with measurable disease at baseline, received at least 1 dose of study medication, and had correct histological cancer type.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 33
percentage of participants | 42.4 [25.5 to 60.8]

5. Secondary Outcome: Ratio to Baseline (Bsl) in Median Levels of Soluble Protein Biomarkers by Prostate Specific Antigen (PSA) Response: VEGFC
Description: Soluble protein biomarker Vascular Endothelial Growth Factor C (VEGFC) measured as picograms per milliliter (pg/mL). PSA responders are participants with a confirmed PSA response as per the Working Group criteria (>50% decrease from baseline) and non-responders are those not meeting the definition of responder. Ratio=value of soluble protein biomarkers at each time point to the value at baseline (C1D14 : C1D1).
Time Frame: Baseline (Cycle 1 Day 1 [C1.D1]), C1.D14, C2.D1, C2.D14, C3.D1, C3.D14
Population: ITT
Measure: Median (Full Range); unit: pg/mL
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 55
pg/mL
  Bsl median - PSA responder | 622.70 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  Bsl median - PSA non-responder | 639.70 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C1D14 : C1D1 - PSA responder | 1.06 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C1D14 : C1D1 - PSA non-responder | 1.07 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D1 : C1D1 - PSA responder | 0.88 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D1 : C1D1 - PSA non-responder | 0.93 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D14 : C1D1 - PSA responder | 0.92 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D14 : C1D1 - PSA non-responder | 0.95 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D1 : C1D1 - PSA responder | 1.51 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D14 : C1D1 - PSA responder | 0.97 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D14 : C1D1 - PSA non-responder | 0.96 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
Statistical Analysis 1: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C1D14 : C1D1; Test type: Superiority or Other; p = 0.942, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C2.D1 : C1D1; Test type: Superiority or Other; p = 0.323, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C2.D14 : C1D1; Test type: Superiority or Other; p = 0.865, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C3.D14 : C1D1; Test type: Superiority or Other; p = 0.873, Wilcoxon rank-sum test

6. Secondary Outcome: Ratio to Baseline in Median Levels of Soluble Protein Biomarkers by Prostate Specific Antigen (PSA) Response: VEGFR2
Description: Soluble protein biomarker Vascular Endothelial Growth Factor receptor 2 (VEGFR2) measured as pg/mL. PSA responders are participants with a confirmed PSA response as per the Working Group criteria (>50% decrease from baseline) and non-responders are those not meeting the definition of responder. Ratio=value of soluble protein biomarkers at each time point to the value at baseline (C1D14 : C1D1).
Time Frame: Baseline (C1.D1), C1.D14, C2.D1, C2.D14, C3.D1, C3.D14
Population: ITT
Measure: Median (Full Range); unit: pg/mL
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 55
pg/mL
  Bsl median - PSA responder | 9889.00 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  Bsl median - PSA non-responder | 10324.00 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C1D14 : C1D1 - PSA responder | 0.73 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C1D14 : C1D1 - PSA non-responder | 0.68 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D1 : C1D1 - PSA responder | 0.80 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D1 : C1D1 - PSA non-responder | 0.79 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D14 : C1D1 - PSA responder | 0.67 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D14 : C1D1 - PSA non-responder | 0.60 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D1 : C1D1 - PSA responder | 0.81 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D14 : C1D1 - PSA responder | 0.63 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D14 : C1D1 - PSA non-responder | 0.67 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
Statistical Analysis 1: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C1D14 : C1D1; Test type: Superiority or Other; p = 0.736, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C2.D1 : C1D1; Test type: Superiority or Other; p = 0.962, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C2.D14 : C1D1; Test type: Superiority or Other; p = 0.185, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C3.D14 : C1D1; Test type: Superiority or Other; p = 1.000, Wilcoxon rank-sum test

7. Secondary Outcome: Ratio to Baseline in Median Levels of Soluble Protein Biomarkers by Prostate Specific Antigen (PSA) Response: VEGFR3
Description: Soluble protein biomarker Vascular Endothelial Growth Factor Receptor 3 (VEGFR3) measured as picograms per milliliter (pg/mL). PSA responders are participants with a confirmed PSA response as per the Working Group criteria (>50% decrease from baseline) and non-responders are those not meeting the definition of responder. Ratio=value of soluble protein biomarkers at each time point to the value at baseline (C1D14 : C1D1).
Time Frame: Baseline (C1.D1), C1.D14, C2.D1, C2.D14, C3.D1, C3.D14
Population: ITT
Measure: Median (Full Range); unit: pg/mL
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 55
pg/mL
  Bsl median - PSA responder | 22475.00 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  Bsl median - PSA non-responder | 22070.00 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C1D14 : C1D1 - PSA responder | 0.69 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C1D14 : C1D1 - PSA non-responder | 0.73 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D1 : C1D1 - PSA responder | 0.75 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D1 : C1D1 - PSA non-responder | 0.75 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D14 : C1D1 - PSA responder | 0.65 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D14 : C1D1 - PSA non-responder | 0.72 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D1 : C1D1 - PSA responder | 0.65 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D14 : C1D1 - PSA responder | 0.56 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D14 : C1D1 - PSA non-responder | 0.66 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
Statistical Analysis 1: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C1D14 : C1D1; Test type: Superiority or Other; p = 0.386, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C2.D1 : C1D1; Test type: Superiority or Other; p = 0.904, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C2.D14 : C1D1; Test type: Superiority or Other; p = 0.812, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C3.D14 : C1D1; Test type: Superiority or Other; p = 0.490, Wilcoxon rank-sum test

8. Secondary Outcome: Ratio to Baseline in Median Levels of Soluble Protein Biomarkers by Clinical Benefit Response (CBR): VEGFC
Description: Soluble protein biomarker VEGFC measured as pg/mL. CBR defined as confirmed CR (disappearance of all target lesions) or confirmed PR (≥30% decrease in sum of longest dimensions [LD] of target lesions taking as reference the baseline sum LD) or SD (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease) ≥3 months versus PD (≥20% increase in sum LD of target lesions taking as reference the smallest sum LD recorded since treatment started, unequivocal progression of existing non-target lesions, or appearance of ≥1 new lesions) or SD <3 months.
Time Frame: Baseline (C1.D1), C1.D14, C2.D1, C2.D14, C3.D14
Population: ITT
Measure: Median (Full Range); unit: pg/mL
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 55
pg/mL
  Bsl median - CR or PR | 581.05 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  Bsl median - SD or PD | 586.85 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C1D14 : C1D1 - CR or PR | 1.21 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C1D14 : C1D1 - SD or PD | 1.19 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D1 : C1D1 - CR or PR | 0.89 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D1 : C1D1 - SD or PD | 1.15 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D14 : C1D1 - CR or PR | 0.92 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D14 : C1D1 - SD or PD | 0.97 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D14 : C1D1 - CR or PR | 0.88 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D14 : C1D1 - SD or PD | 0.59 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
Statistical Analysis 1: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C1D14 : C1D1; Test type: Superiority or Other; p = 0.839, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C2.D1 : C1D1; Test type: Superiority or Other; p = 0.219, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C2.D14 : C1D1; Test type: Superiority or Other; p = 0.788, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C3.D14 : C1D1; Test type: Superiority or Other; p = 0.164, Wilcoxon rank-sum test

9. Secondary Outcome: Ratio to Baseline in Median Levels of Soluble Protein Biomarkers by Clinical Benefit Response (CBR): VEGFR2
Description: Soluble protein biomarker VEGFR2 measured as pg/mL. CBR defined as confirmed CR (disappearance of all target lesions) or confirmed PR (≥30% decrease in sum of longest dimensions [LD] of target lesions taking as reference the baseline sum LD) or SD (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease) ≥3 months versus PD (≥20% increase in sum LD of target lesions taking as reference the smallest sum LD recorded since treatment started, unequivocal progression of existing non-target lesions, or appearance of ≥1 new lesions) or SD <3 months.
Time Frame: Baseline (C1.D1), C1.D14, C2.D1, C2.D14, C3.D14
Population: ITT
Measure: Median (Full Range); unit: pg/mL
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 55
pg/mL
  Bsl median - CR or PR | 9837.50 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  Bsl median - SD or PD | 9484.25 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C1D14 : C1D1 - CR or PR | 0.73 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C1D14 : C1D1 - SD or PD | 0.75 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D1 : C1D1 - CR or PR | 0.83 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D1 : C1D1 - SD or PD | 0.83 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D14 : C1D1 - CR or PR | 0.68 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D14 : C1D1 - SD or PD | 0.60 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D14 : C1D1 - CR or PR | 0.63 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D14 : C1D1 - SD or PD | 0.80 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
Statistical Analysis 1: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C1D14 : C1D1; Test type: Superiority or Other; p = 0.656, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C2.D1 : C1D1; Test type: Superiority or Other; p = 0.628, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C2.D14 : C1D1; Test type: Superiority or Other; p = 0.420, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C3.D14 : C1D1; Test type: Superiority or Other; p = 0.296, Wilcoxon rank-sum test

10. Secondary Outcome: Ratio to Baseline in Median Levels of Soluble Protein Biomarkers by Clinical Benefit Response (CBR): VEGFR3
Description: Soluble protein biomarker VEGFR3 measured as pg/mL. CBR defined as confirmed CR (disappearance of all target lesions) or confirmed PR (≥30% decrease in sum of longest dimensions [LD] of target lesions taking as reference the baseline sum LD) or SD (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease) ≥3 months versus PD (≥20% increase in sum LD of target lesions taking as reference the smallest sum LD recorded since treatment started, unequivocal progression of existing non-target lesions, or appearance of ≥1 new lesions) or SD <3 months.
Time Frame: Baseline (C1.D1), C1.D14, C2.D1, C2.D14, C3.D14
Population: ITT
Measure: Median (Full Range); unit: pg/mL
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 55
pg/mL
  Bsl median - CR or PR | 19975.00 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  Bsl median - SD or PD | 22495.00 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C1D14 : C1D1 - CR or PR | 0.72 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C1D14 : C1D1 - SD or PD | 0.68 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D1 : C1D1 - CR or PR | 0.78 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D1 : C1D1 - SD or PD | 0.83 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D14 : C1D1 - CR or PR | 0.69 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C2.D14 : C1D1 - SD or PD | 0.80 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D14 : C1D1 - CR or PR | 0.61 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
  C3.D14 : C1D1 - SD or PD | 0.78 [NA to NA] — Measure of dispersion was not calculated for the median; the data was not mature.
Statistical Analysis 1: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C1D14 : C1D1; Test type: Superiority or Other; p = 0.903, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C2.D1 : C1D1; Test type: Superiority or Other; p = 0.434, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C2.D14 : C1D1; Test type: Superiority or Other; p = 0.687, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg; C3.D14 : C1D1; Test type: Superiority or Other; p = 0.296, Wilcoxon rank-sum test

11. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory-Short Form (mBPI-sf) : Pain Intensity (Questions 2-5)
Description: The questionnaire assesses pain intensity (worst, least, average, and right now), level of relief in the last 24 hours, and the impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life). The pain intensity index score was derived from Questions 2-5 with range from 0 to 10 (0: no pain; 1-4: mild pain; 5-6: moderate pain; 7-10: severe pain); higher scores indicate worse health status.
Time Frame: Baseline (C1.D1), Day 1 of Cycles 2 through 16, and End of Treatment (EOT=following Cycle 16 or within 7 days of withdrawal from study)
Population: Patient reported outcomes (PRO) evaluable population defined as participants in the ITT population who received at least 1 dose of study medication (sunitinib or docetaxel) and had baseline data; (n)=number of participants with evaluable data at observation.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 48
scores on a scale
  Bsl mean C1.D1 (n=48) | 1.9 [1.4 to 2.4]
  Change from Bsl - C2.D1 (n=42) | -1.0 [-1.4 to -0.5]
  Change from Bsl - C3.D1 (n=35) | -1.1 [-1.7 to -0.5]
  Change from Bsl - C4.D1 (n=30) | -0.8 [-1.7 to 0.0]
  Change from Bsl - C5.D1 (n=32) | -0.8 [-1.7 to 0.1]
  Change from Bsl - C6.D1 (n=32) | -0.8 [-1.6 to 0.0]
  Change from Bsl - C7.D1 (n=29) | -0.8 [-1.6 to -0.1]
  Change from Bsl - C8.D1 (n=26) | -0.7 [-1.7 to 0.3]
  Change from Bsl - C9.D1 (n=25) | -0.5 [-1.3 to 0.4]
  Change from Bsl - C10.D1 (n=22) | -0.7 [-1.5 to 0.0]
  Change from Bsl - C11.D1 (n=21) | -1.2 [-2.0 to -0.5]
  Change from Bsl - C12.D1 (n=18) | -0.8 [-1.8 to 0.1]
  Change from Bsl - C13.D1 (n=17) | -1.2 [-2.1 to -0.3]
  Change from Bsl - C14.D1 (n=17) | -1.3 [-2.1 to -0.6]
  Change from Bsl - C15.D1 (n=12) | -1.1 [-2.2 to 0.1]
  Change from Bsl - C16.D1 (n=12) | -0.5 [-2.6 to 1.6]
  Change from Bsl - EOT (n=37) | -0.3 [-1.0 to 0.3]

12. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory-Short Form (mBPI-sf): Pain Interference (Questions 7A Through 7G)
Description: The questionnaire assesses pain intensity (worst, least, average, and right now), level of relief in the last 24 hours, and the impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life). The pain interference index score (to measure how much pain had interfered with daily activities) was derived from Questions 7A-7G with a range from 0 (no interference) to 10 (completely interferes); higher scores indicate more interference.
Time Frame: as for outcome 11
Population: PRO evaluable population; (n)=number of participants with evaluable data at observation.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 48
scores on a scale
  Bsl mean C1.D1 (n=48) | 1.8 [1.2 to 2.4]
  Change from Bsl - C2.D1 (n=41) | -0.7 [-1.1 to -0.3]
  Change from Bsl - C3.D1 (n=34) | -0.8 [-1.5 to -0.2]
  Change from Bsl - C4.D1 (n=30) | -0.5 [-1.4 to 0.5]
  Change from Bsl - C5.D1 (n=31) | -0.7 [-1.8 to 0.4]
  Change from Bsl - C6.D1 (n=32) | -0.6 [-1.4 to 0.3]
  Change from Bsl - C7.D1 (n=29) | -0.4 [-1.1 to 0.4]
  Change from Bsl - C8.D1 (n=26) | -0.5 [-1.3 to 0.3]
  Change from Bsl - C9.D1 (n=24) | -0.5 [-1.3 to 0.3]
  Change from Bsl - C10.D1 (n=21) | -0.4 [-1.3 to 0.5]
  Change from Bsl - C11.D1 (n=21) | -0.7 [-1.7 to 0.3]
  Change from Bsl - C12.D1 (n=18) | -0.8 [-2.0 to 0.4]
  Change from Bsl - C13.D1 (n=17) | -1.2 [-2.2 to -0.1]
  Change from Bsl - C14.D1 (n=17) | -1.4 [-2.3 to -0.5]
  Change from Bsl - C15.D1 (n=12) | -1.0 [-2.0 to 0.1]
  Change from Bsl - C16.D1 (n=12) | -0.5 [-2.1 to 1.1]
  Change from Bsl - EOT (n=36) | -0.4 [-1.1 to 0.2]

13. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Prostate (FACT-P) Questionnaire (FACT-General and Prostate Cancer Subscale)
Description: Assesses health related quality of life and advanced prostate cancer specific symptoms. FACT-General (FACT-G) assesses 4 domains: physical, social and family, emotional, and functional well-being. The prostate cancer subscale assesses prostate cancer symptoms focusing on pain, urination problems, and sexual functions. Individual scores range from 0 (not at all) to 4 (very much). Scores for some of the individual questions are reverse-coded in order for higher scores to correspond to better health status. FACT-P overall score range is 0 to 156; higher scores indicate better health status.
Time Frame: as for outcome 11
Population: PRO evaluable population; (n)=number of participants with evaluable data at observation.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 48
scores on a scale
  Bsl mean C1.D1 (n=47) | 112.0 [107.0 to 117.0]
  Change from Bsl - C2.D1 (n=42) | 6.4 [2.2 to 10.6]
  Change from Bsl - C3.D1 (n=31) | 7.2 [3.5 to 11.0]
  Change from Bsl - C4.D1 (n=30) | 6.6 [0.2 to 13.0]
  Change from Bsl - C5.D1 (n=33) | 4.9 [-1.5 to 11.4]
  Change from Bsl - C6.D1 (n=31) | 8.2 [3.4 to 13.0]
  Change from Bsl - C7.D1 (n=29) | 4.4 [-0.4 to 9.1]
  Change from Bsl - C8.D1 (n=25) | 3.6 [-1.8 to 9.0]
  Change from Bsl - C9.D1 (n=24) | 0.2 [-5.0 to 5.4]
  Change from Bsl - C10.D1 (n=22) | 2.0 [-4.8 to 8.8]
  Change from Bsl - C11.D1 (n=21) | 3.1 [-3.9 to 10.1]
  Change from Bsl - C12.D1 (n=18) | 4.1 [-2.5 to 10.7]
  Change from Bsl - C13.D1 (n=16) | 5.6 [-2.2 to 13.5]
  Change from Bsl - C14.D1 (n=17) | 7.9 [0.6 to 15.2]
  Change from Bsl - C15.D1 (n=12) | 4.1 [-2.5 to 10.7]
  Change from Bsl - C16.D1 (n=12) | 6.2 [-1.9 to 14.2]
  Change from Bsl - EOT (n=36) | 0.6 [-4.5 to 5.8]

14. Secondary Outcome: Preliminary Assessment of PSA Modulation by SU011248
Description: PSA modulation analyzed by the mean change in PSA response measured as ng/mL.
Time Frame: Baseline to Day 28
Population: ITT population; PSA modulation was listed as a secondary endpoint for Phase 2, however, modulation was planned for analysis only for Phase 1 portion of the study. No formal analysis was completed to determine modulation.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg
Serious Adverse Events (participants affected / at risk) | 28/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg (N=55)
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Arrhythmia supraventricular (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 2
Mucosal inflammation (General disorders) | 1
Multi-organ failure (General disorders) | 1
Pyrexia (General disorders) | 2
Cholestasis (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pseudomonas infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Transaminases increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Haematoma (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SU011248 37.5 mg + Docetaxel 75 mg/m^2 + Prednisone 5 mg (N=55)
Anaemia (Blood and lymphatic system disorders) | 17
Leukopenia (Blood and lymphatic system disorders) | 23
Lymphopenia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 33
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Lacrimation increased (Eye disorders) | 16
Abdominal pain (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 44
Dry mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 12
Dysphagia (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7
Gingivitis (Gastrointestinal disorders) | 3
Glossodynia (Gastrointestinal disorders) | 10
Haemorrhoids (Gastrointestinal disorders) | 3
Mouth ulceration (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 33
Oral pain (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 20
Asthenia (General disorders) | 8
Chest pain (General disorders) | 7
Chills (General disorders) | 7
Fatigue (General disorders) | 44
Influenza like illness (General disorders) | 6
Mucosal inflammation (General disorders) | 20
Oedema peripheral (General disorders) | 20
Pain (General disorders) | 6
Pyrexia (General disorders) | 15
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Bronchitis (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 3
Tooth abscess (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 7
Contusion (Injury, poisoning and procedural complications) | 7
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 6
Blood creatinine increased (Investigations) | 6
Haemoglobin decreased (Investigations) | 4
Weight decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 14
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 19
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14
Hypocalcaemia (Metabolism and nutrition disorders) | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Dizziness (Nervous system disorders) | 13
Dysgeusia (Nervous system disorders) | 34
Headache (Nervous system disorders) | 8
Hypoaesthesia (Nervous system disorders) | 4
Neuropathy peripheral (Nervous system disorders) | 13
Peripheral sensory neuropathy (Nervous system disorders) | 7
Tremor (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 3
Dysuria (Renal and urinary disorders) | 11
Haematuria (Renal and urinary disorders) | 4
Incontinence (Renal and urinary disorders) | 4
Nocturia (Renal and urinary disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 35
Dry skin (Skin and subcutaneous tissue disorders) | 12
Hair colour changes (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 14
Night sweats (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 15
Rash (Skin and subcutaneous tissue disorders) | 15
Skin depigmentation (Skin and subcutaneous tissue disorders) | 3
Skin discolouration (Skin and subcutaneous tissue disorders) | 8
Swelling face (Skin and subcutaneous tissue disorders) | 4
Sinus operation (Surgical and medical procedures) | 3
Flushing (Vascular disorders) | 4
Haematoma (Vascular disorders) | 3
Hot flush (Vascular disorders) | 3
Hypertension (Vascular disorders) | 7
Deep vein thrombosis (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
Per FDAAA, only the Phase 2 study results are posted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.